CLINICAL TRIAL: NCT01593332
Title: Low Dose Rituximab as a First Line Biologic Therapy for the Treatment of DMARD Resistant Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Kamila Hashemzadeh, assisstant professor, Mashhad University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 87549; 87549 (Other: DEPUTY OF RESEARCH OF MASHHAD UNIVERSITY OF MEDICAL SCIENCES)
Record Dates: First submitted 2012-01-07; First posted 2012-05-08 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: DMARD Resistant Rheumatoid Arthritis
Keywords: Rituximab; Rheumatoid arthritis; Biologics; Anti-tumour necrosis factor; Disease-modifying anti-rheumatic drugs; DAS28; European League Against Rheumatism response
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab (Active Comparator)
  Interventions: Drug: Rituximab
- Methotrexate (Active Comparator)
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — two 500 mg rituximab infusions 2 weeks apart
  Other Names: Mabthera
Drug: Rituximab — 500mg,two times with two weeks interval
  Other Names: Mabthera

SUMMARY:
In this project the investigators decide to evaluate the efficacy and safety of half dose mabthera (it means 500 mg infusion two weeks apart) in conventional drug resistant cases of rheumatoid arthritis. The investigators choose this drug because the use of anti-TNF drugs limited in the investigators refractory patients as the first line drugs because of its cost.

ELIGIBILITY:
Inclusion Criteria:

* 1987 ACR criteria for classification of RA
* Positive for rheumatoid factor(RF)
* Active RA despite therapy with conventional for at least 3 months as evidenced by DAS 28 > 3/2
* Patients with active, resistant RA who didn't receive anti TNF agents.

Exclusion Criteria:

* Patient with hypogammaglobulinemia
* Patient with congestive heart failure (classIV)
* Active current bacterial,viral,fungal,myocardial or other infections
* Chronic hepatitis B or hepatitis C carriers
* History of severe allergic reaction to human,humanized or murine monoclonal antibodies
* History of malignancies
* Pregnant women or lactating mothers 8) Patients with Chronic renal failure and hepatic disease.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-07; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
change in 28-joint disease activity index( DAS28) | Study duration was 6 months and the subjects were assessed for DAS 28 change at baseline, after 2 , 16 and 24 weeks.
  disease activity score 28 formula which caculates based the number of tenderness and swelling of 28 joints and also ESR)
Change in European league against rheumatism(EULAR) response criteria | Change in EULAR 2,16,24 weeks

SECONDARY OUTCOMES:
Rituximab side effects | 0,2,16,24 weeks
  side effects like infusion reaction , paresthesia, itching,hypertension or hypotension,headache and infection.

CONTACTS AND LOCATIONS:
Locations (1):
- Rheumatic Diseases Research Center, Mashhad University of Medical Sciences, Mashhad, Khorasan Razavi, Iran